CLINICAL TRIAL: NCT05955898
Title: The Development and Evaluation of a Single Session Intervention for Parent Distress Tolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, Associate Chair, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230552
Record Dates: First submitted 2023-06-18; First posted 2023-07-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-09

CONDITIONS: Parents; Mental Health Issue; Distress, Emotional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parents THRIVE Group (Experimental): Participants in this group will receive the Parents THRIVE intervention. Participants will be in this group for up to two hours.
  Interventions: Behavioral: Parents THRIVE
- Sharing Feelings Project Group (Active Comparator): Participants in this group will receive the Sharing Feelings Group intervention. Participants will be in this group for up to two hours.
  Interventions: Behavioral: Sharing Feelings Project

INTERVENTIONS:
Behavioral: Parents THRIVE — Parents THRIVE is a digital, one-time intervention that will give parents strategies to cope with their emotions and improve their distress tolerance. Parents will learn how to increase their emotion awareness to better tolerate strong emotions, such as anxiety, sadness, anger, and frustration.
  Arms: Parents THRIVE Group
Behavioral: Sharing Feelings Project — Sharing Feelings Project is a digital, one-time program that focuses on the benefit of sharing emotions with others and will be used as a control. Parents will read about how sharing their emotions can be helpful and anecdotes from others' experiences sharing emotions.
  Arms: Sharing Feelings Project Group

SUMMARY:
The purpose of this study is to study different ways to help parents cope with strong emotions. The study team will be looking at how two different treatments help parents learn to manage strong emotions. These treatments are one session and are completed online, without a therapist, like an online training or class.

ELIGIBILITY:
Inclusion Criteria:

* Live in the United States.
* Parent of a child aged 6-17 years old who has received at least one counseling or mental health treatment session from a provider in the last 6 months will be eligible to participate.
* Parent is not currently receiving psychotherapy or counseling for a mental health concern (or received such in the past six months).
* Parent reported poor distress tolerance (DT). Poor DT will be defined as a score of less than 54 on the Distress Tolerance Scale.
* Due to language limitations of the primary researcher, parents will be eligible if they comfortably speak and read in English.
* Parents must have a mobile device (e.g., laptop, tablet, smart phone, etc.) or desktop computer and internet access sufficient for the delivery of the study assessments and intervention online.

Exclusion Criteria:

* Failure to meet any of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Change in Distress Tolerance Scale scores | Baseline, up to three-week follow-up
  The Distress Tolerance Scale is a 15-item self-report measure that measures the perceived capacity to tolerate distress from a multidimensional framework, including tolerance, appraisal, absorption, and regulation. Items are rated on a 1-5 Likert scale and then summed. Scores range from 15-75. Higher total scores indicate greater ability to tolerate distress.

SECONDARY OUTCOMES:
Change in Overall Anxiety Severity and Impairment Scale (OASIS) scores | Baseline, up to three-week follow-up
  Measures overall anxiety severity and anxiety-related impairment due to any anxiety disorder. Total scores are computed by summing scores from all 5 items. Total score ranges from 0 to 20, with higher scores indicating higher severity and impairment of anxiety symptoms. Reduction in OASIS scores therefore indicates better outcome.
Change in Overall Depression Severity and Impairment Scale (ODSIS) scores | Baseline, up to three-week follow-up
  Measures severity and frequency of depressive symptoms and functional deficits in pleasurable activities due to the depressive symptomatology. The ODSIS consists of 5 self-report items rated from 0 to 4. Total score ranges from 0 to 20 with higher scores indicating greater depression-related severity and impairment.
Change in Parental Acceptance and Action Questionnaire (PAAQ) scores | Baseline, up to three-week follow-up
  A 19-item measure of parent experiential avoidance, or parental actions intended to control the form and frequency of their child's emotional experiences. Items are rated on a 7-point scale, with higher possible scores ranging from 19 to 133. Higher scores indicate less parental experiential avoidance and less effort to control child emotional experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami; Elizabeth R Halliday, MS, Study Chair — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheron DM, Ehrenreich JT, Pincus DB. Assessment of parental experiential avoidance in a clinical sample of children with anxiety disorders. Child Psychiatry Hum Dev. 2009 Sep;40(3):383-403. doi: 10.1007/s10578-009-0135-z. Epub 2009 Mar 12. PMID 19280337
- [Background] Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. Motivation and Emotion, 29(2), 83-102.
- [Background] Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-9. doi: 10.1002/da.20182. PMID 16688739
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Schleider, J. L., & Weisz, J. R. (2019). Sharing feelings project. Open Science Framework.
- [Background] Schleider JL, Dobias ML, Sung JY, Mullarkey MC. Future Directions in Single-Session Youth Mental Health Interventions. J Clin Child Adolesc Psychol. 2020 Mar-Apr;49(2):264-278. doi: 10.1080/15374416.2019.1683852. Epub 2019 Dec 4. PMID 31799863
- [Background] Ehrenreich-May, J., Kennedy, S. M., Sherman, J. A., Bilek, E. L., Buzzella, B. A., Bennett, S. M., & Barlow, D. H. (2017). Unified protocols for transdiagnostic treatment of emotional disorders in children and adolescents: Therapist guide. Oxford University Press.
- [Background] Barlow, D. H., Farchione, T. J., Sauer-Zavala, S., Latin, H. M., Ellard, K. K., Bullis, J. R., ... & Cassiello-Robbins, C. (2017). Unified protocol for transdiagnostic treatment of emotional disorders: Therapist guide. Oxford University Press.